CLINICAL TRIAL: NCT01302574
Title: The Role of Sweet Taste Receptor Blockade on Intragastric Liquid Meal-stimulated Secretion of Satiation Peptides in Healthy Humans
Brief Title: Role of the Gut Sweet Taste Receptor in the Secretion of Satiation Peptides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Beglinger Christoph, Prof. Dr. med., Department of Gastroenterology, University Hospital Basel, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 69/04.02
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Taste Disorder, Secondary, Sweet
Keywords: T1R2/T1R3; gastric emptying; gut; lactisole; nutrient sensing
MeSH Terms: conditions — Taste Disorders | interventions — lactisole; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mixed liquid meal (Placebo Comparator): 500 mL mixed liquid meal + 50 mg 13C-sodium-acetate
  Interventions: Dietary Supplement: lactisole
- mixed liquid meal + lactisole (Active Comparator): 500 mL mixed liquid meal + 50 mg 13C-sodium-acetate + 450 ppm lactisole
  Interventions: Dietary Supplement: lactisole

INTERVENTIONS:
Dietary Supplement: lactisole — Lactisole-liquid meal: Lactisole (450 ppm) will be mixed with a liquid meal. Liquid meal only: The comparator will be the liquid meal alone.
  Other Names: Dietary supplement

SUMMARY:
The purpose of this study is to determine the functional significance of sweet taste receptors in the secretion of gastrointestinal (GI) satiation peptides by using a specific sweet taste receptor antagonist to block sweet taste perception in the gastrointestinal tract.

DETAILED DESCRIPTION:
There is strong evidence that taste signaling mechanisms identified in the oral epithelium also operate in the gut. It is suggested that open-type enteroendocrine cells directly sense nutrient via alpha-gustducin coupled taste receptors to modulate the secretion of glucagon like peptide-1 (GLP-1) and peptide YY (PYY). Several nutrient responsive G-protein coupled receptors have been identified in the human gut, including the sweet taste responsive T1R2/T1R3 heterodimer, the amino acid/umami responsive T1R1/T1R3 as well as GPR120 for unsaturated long-chain free fatty acids. The functional significance of sweet taste receptors in mixed liquid meal-stimulated secretion of GLP-1 and PYY will be determined by intragastric infusion of a 500 mL mixed liquid meal with or without lactisole (450 ppm)in a double blind, 2-way crossover trial including 16 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* BMI of 19.0-24.5
* age 18-40 years old
* stable body weight for at least 3 month

Exclusion Criteria:

* smoking
* substance abuse
* regular intake of medication
* medical or psychiatric illness
* gastrointestinal disorders or food allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal peptide secretion | 2 hours blood sampling

SECONDARY OUTCOMES:
Appetite perceptions | 4 hours
Gastric emptying rate | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Phase 1 Research Unit, University Hospital Basel
Locations (1):
- University Hospital Basel, Phase 1 Research Unit, Basel, Switzerland